CLINICAL TRIAL: NCT01765257
Title: Evaluation of the Efficacy of Rasagiline in Apathy in Drug-naïve Patients With Parkinson's Disease by a Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled Study.
Brief Title: Evaluation of the Efficacy of Rasagiline in Apathy in Drug-naïve Patients With Parkinson's Disease by a Multi-center Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: H. Lundbeck A/S (Industry); CHU Purpan (Toulouse) (Unknown); Hôpital Haut-Lévêque (Other); Centre Hospitalier de la côte Basque (Other); Poitiers University Hospital (Other); CHU de Rennes (Rennes) (Unknown); University Hospital, Lille (Other); Hôpital Dupuytren (Other); University Hospital, Caen (Other); Centre Hospitalier Universitaire de Nīmes (Other); Centre Hospitalier du Pays d'Aix (Other); Hôpital de la Timone (MARSEILLE) (Unknown); University Hospital, Rouen (Other); Centre Hospitalier Universitaire, Amiens (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Fondation Rothschild Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0138; 2007-002800-16
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Drug-naïve Patients With Parkinson's Disease; Apathy
Keywords: Drug-naïve patients with Parkinson's disease; Apathy; Rasagiline
MeSH Terms: conditions — Lethargy | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- rasagiline (Experimental): Randomized, double-blind, rasagiline (1 mg) vs placebo study. Parallel group (randomization 1/1). Duration 3 months 16 recruiting centers in France
  Interventions: Drug: AZILECT®
- placebo (Placebo Comparator): Randomized, double-blind, rasagiline (1 mg) vs placebo study. Parallel group (randomization 1/1). Duration 3 months 16 recruiting centers in France
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZILECT®
  Arms: rasagiline
Drug: Placebo
  Arms: placebo

SUMMARY:
Among the psychiatric symptoms observed in the premotor phase of Parkinson's disease (PD) and/or in "de novo" patients, apathy is relatively frequent (estimated to 23%). However, the neuropathological bases of apathy are still unknown. However, recent data suggests that apathy could be linked to a more specific dopaminergic denervation in the ventral striatum.

Rasagiline increases the bioavailability of striatal endogenous dopamine by blocking the MAO-B. Some recent data suggest rasagiline could be effective to improve apathy in Parkinson's disease.

The primary outcome is to demonstrate a significant reduction of apathy using the Lille apathy rating scale (LARS) in drug naive patients with early diagnosed Parkinson's disease, using a treatment by rasagiline.

DETAILED DESCRIPTION:
Study design :

Randomized, double-blind, rasagiline (1 mg) vs placebo study. Parallel group (randomization 1/1). Duration 3 months 16 recruiting centers in France

Population :

50 drug-naïve patients with Parkinson's disease, with apathy. 2 groups : 25 patients with placebo and 25 patients with rasagiline.

3 visits

* Visit 1 : inclusion / randomisation/ first study medication dispensation
* Visit 2 (1.5 month after V1) : first evaluation and second study medication dispensation.
* Visit 3 (3 months after V1, final visit) : second evaluation

ELIGIBILITY:
Inclusion Criteria:

- Drug-naïve patients with Parkinson's disease (UKPDBB criteria)

* No dementia (Mattis dementia rating scale > 130; Mini Mental Sate Examination ≥26)
* No depression (MADRS < 15)
* Criteria of apathy from Robert et al (2009)
* At least mild apathy (≥-21 to Lille Apathy Rating Scale)
* Age : 35-70 y
* Affiliation to social security
* Agreement of patients

Exclusion Criteria:

* - Any antiparkinsonian treatment (L.dopa, dopamine agonists, MAO-B-I, amantadine, anticholinergics). Patients treated by dopamine agonists but who have stopped it more than 3 months before their inclusion can be included.
* Ongoing severe psychiatric or somatic diseases
* Others treatments :
* antipsychotics
* antidepressants and anxiolytics (exclusion if the treatment is not stable the month before inclusion)
* psychostimulants (methylphenidate, adrafinil, modafinil, deanol, vitamin C, sulbutiamine, glutamic acid, aspartic acid)
* any contra-indication according to SmPC
* patients under guardianship
* Women without efficient contraception
* Person who participate to an other study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Lille Apathy Rating Scale (LARS) score | at the visit 3 (after 3 months of treatment)

SECONDARY OUTCOMES:
Motor assessment : Unified Parkinson's Disease Rating Scale | at the visit 3 (after 3 months of treatment)
Depressive and anxiety symptoms : MADRS + Hamilton anxiety scale | at the visit 3 (after 3 months of treatment)
Self assessment of apathy : Starkstein | at the visit 3 (after 3 months of treatment)
Quality of life : PDQ 39 | at the visit 3 (after 3 months of treatment)
Cognitive assessment: MATTIS dementia rating scale, MMSE, executive functions battery | at the visit 3 (after 3 months of treatment)
Hyperdopaminergic symptoms : Parkinson's disease behavioral scale | at the visit 3 (after 3 months of treatment)
Fatigue assessment : Parkinson Fatigue Scale | at the visit 3 (after 3 months of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Denis PEZET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France